CLINICAL TRIAL: NCT03921723
Title: Non-randomized, Sequential, Fixed-sequence Evaluation of Prototype Dolutegravir Liquid Formulations Versus 5mg Dolutegravir Dispersible Tablets Following Single-dose Fasted-state Administrations to Normal Healthy Adult Participants
Brief Title: Dolutegravir Pediatric Liquid Formulation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 209354
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: Dolutegravir; Human immunodeficiency virus; Sequential study; Dispersible tablet; Suspension; Liquid solution
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: The study is non-randomized 6 period, 6 way fixed sequential design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subject receiving Dolutegravir 10 mg (Experimental): Subject will receive a prototype equivalent to DTG 10 mg liquid formulation in period 1, a prototype equivalent to DTG 10 mg liquid formulation in period 2, a DTG 10 mg dispersible tablet in Period 3, each period will be separated by washout period of >= 7 days, if required a prototype equivalent to DTG 10 mg liquid formulation in period 4, a prototype equivalent to DTG 10 mg liquid formulation in period 5, and a prototype equivalent to DTG 10 mg liquid formulation in period 6 will be evaluated.
  Interventions: Drug: Dolutegravir dispersible tablet; Drug: Dolutegravir oral suspension; Drug: Dolutegravir oral solution

INTERVENTIONS:
Drug: Dolutegravir dispersible tablet — DTG will be available as an oral tablet with dosing strength of 5 mg 2 tablet will be dispersed in water will be administered orally for prescribed regimen.
Drug: Dolutegravir oral suspension — DTG will be available as an oral suspension with dosing strength of 5 mg per milliliter (ml) or 2 mg per ml with miglyol 812N or ethyl cellulose in miglyol 812N as vehicle for suspension administered orally for prescribed regimen.
Drug: Dolutegravir oral solution — DTG will be available as an oral solution with dosing strength of 2 mg per ml will be administered orally for prescribed regimen.

SUMMARY:
This is an open-label, single-center, single dose, non-randomized, sequential, fixed-sequence study, which will evaluate pharmacokinetics (PK) of dolutegravir (DTG) in healthy adult subjects. The study will contain 6 periods with five prototype liquid formulations for evaluation in fasted state. In period 1, 2 and 3 single reference dose of 2 dispersible tablets of 5 milligram DTG will be administered and at least 2 liquid prototype DTG formulations (containing a target total dose of 10mg DTG). There will be a wash-out period of 7 days between each period. In period 4 through 6, there would be options to evaluate additional prototype liquid formulations. The total duration of study will be up to 17 weeks. DTG has been found to be safe and effective in adults infected with human immunodeficiency virus (HIV). DTG dispersible tablets have been developed primarily for use in children from 4 weeks to 6 years of age, and a DTG liquid formulation are is being developed to study the appropriate dose needed for the HIV-exposed and infected neonatal population in the first four weeks of life. Approximately 18 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac evaluation.
* Body weight >= 50 kg (110 pounds [lbs]) for men and >=45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kilogram per meter square (kg/m^2) (inclusive).
* Male and female subjects will be part of study. A female subject is eligible to participate if she is not pregnant or breastfeeding, and is not a woman of childbearing potential (WOCBP).
* Additional requirements for pregnancy testing, if needed, during and after study intervention; The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Subject should be capable of giving signed informed consent as which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigator.
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT correction using Fridericia Formula (QTcF) >450 millisecond (msec)
* Past or intended use of over-the-counter or prescription medication (including herbal medications) within 7 days prior to dosing. Paracetamol.
* History of allergy or sensitivity to DTG.
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation within the last 30 days before signing of consent in this or any other clinical study involving an investigational study intervention or any other type of medical research.
* Presence of Hepatitis B surface antigen (HBsAg), or a positive hepatitis B core antibody with a negative hepatitis B surface antibody at screening.
* Positive Hepatitis C antibody test result at screening: Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) test is obtained.
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* Positive pre-study drug/alcohol screen.
* Positive HIV antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within one month prior to the study defined as: For the United Kingdom an average weekly intake of >14 units for males or females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1, open-label, non-randomized, single dose study in healthy adult participants conducted at a single center in the United Kingdom (UK) to assess the prototype liquid fomulations of dolutegravir (DTG) versus DTG dispersible tablets (reference).
Pre-assignment Details: A total of 22 participants were enrolled in the study. The washout time between dosing in consecutive study periods was a minimum of 7 days.
Groups:
- Prototype A/DTG Reference/Prototype B: Participants were administered a single oral dose of 5 milligrams (mg) per milliliter (mL) DTG sodium oral suspension (Prototype A), for a total of 10 mg in Period 1 followed by a single oral dose of two 5 mg DTG dispersible tablets dispersed in water (DTG reference) in Period 2. Participants further received a single oral dose of 2 mg/mL DTG sodium oral liquid (Prototype B) in Period 3, also receiving a total dose of 10 mg. There was a minimum washout of 7 days between doses.
Period: Period 1 (4 Days)
Arm/Group | Prototype A/DTG Reference/Prototype B
Started | 22
Completed | 22
Not Completed | 0
Period: Period 2 (4 Days)
Arm/Group | Prototype A/DTG Reference/Prototype B
Started | 22
Completed | 19
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Period 3 (4 Days)
Arm/Group | Prototype A/DTG Reference/Prototype B
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prototype A/DTG Reference/Prototype B
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.3 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  CENTRAL/SOUTH ASIAN HERITAGE | 1
  BLACK OR AFRICAN AMERICAN | 2
  WHITE/CAUCASIAN/EUROPEAN HERITAGE | 19

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Time Point (AUC[0-t]) for DTG
Description: Blood samples were collected at indicated time points and pharmacokinetic (PK) analysis was performed. PK parameters were determined by non-compartmental methods.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population comprised of participants in the 'All Participants' (who were randomized and received at least one dose of study medication)' population for whom a PK sample was obtained and had evaluable PK assay results. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Prototype A: Participants received a single oral dose of Prototype A (5 mg/mL DTG oral suspension)
- Prototype B: Participants received a single oral dose of Prototype B (2 mg/mL DTG [as DTG Sodium in glycerol vehicle] oral liquid)
- DTG Reference: Participants received a single oral dose of DTG reference tablets (2x5 mg DTG dispersible tablets dispersed in water)
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours*micrograms per milliliter | 11.9968 (22.7) | 13.7921 (20.5) | 12.1944 (22.7)
Statistical Analysis 1: Comparison: Prototype A vs DTG Reference; Test type: Equivalence — Bioequivalence is established when the 90 percent (%) confidence interval of the ratio for AUC (0 to t) between treatment formulations (Prototype A versus DTG Reference Treatment) are within the range of 0.80 to 1.25; Ratio = 0.97, 90% CI 2-sided [0.91 to 1.03]
Statistical Analysis 2: Comparison: Prototype B vs DTG Reference; Test type: Equivalence — Bioequivalence is established when the 90% confidence interval of the ratio for AUC (0 to t) between treatment formulations (Prototype B versus DTG Reference Treatment) are within the range of 0.80 to 1.25; Ratio = 1.12, 90% CI 2-sided [1.05 to 1.20]

2. Secondary Outcome: Absorption Lag Time (Tlag) Following Administration of DTG
Description: Blood samples were collected at indicated time points and PK analysis was performed. PK parameters were determined by non-compartmental methods.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 0]

3. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours | 1.50 [0.5 to 3.5] | 0.50 [0.5 to 2.0] | 0.75 [0.5 to 5.0]

4. Secondary Outcome: Time of Last Quantifiable Concentration (Tlast) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours | 48.0000 [47.983 to 72.283] | 48.0333 [48.000 to 72.317] | 48.0000 [47.783 to 72.150]

5. Secondary Outcome: Elimination Half-life (t½) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours | 13.6389 (17.5) | 14.5997 (19.1) | 13.5807 (20.9)

6. Secondary Outcome: Apparent Elimination Rate Constant (Lambda z) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Per hour | 0.0508 (17.5) | 0.0475 (19.1) | 0.0510 (20.9)

7. Secondary Outcome: Percentage of AUC(0-inf) Extrapolated (%AUCex) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Percentage of AUCex | 6.1049 (36.8) | 5.8582 (57.1) | 6.3086 (36.3)

8. Secondary Outcome: AUC From Time Zero to 24 Hours (AUC[0-24]) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours*micrograms per milliliter | 9.2541 (16.4) | 10.2918 (15.8) | 9.2356 (18.7)

9. Secondary Outcome: AUC From Time Zero to 72 Hours (AUC[0-72]) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours*micrograms per milliliter | 12.2645 (22.0) | 14.1062 (20.8) | 12.5289 (21.9)

10. Secondary Outcome: Apparent Oral Clearance (CL/F) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Liters per hour | 0.7794 (23.0) | 0.6752 (21.8) | 0.7650 (23.8)

11. Secondary Outcome: Last Quantifiable Concentration (Ct) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Micrograms per milliliter | 0.0398 (35.4) | 0.0412 (53.2) | 0.0421 (39.9)

12. Secondary Outcome: Apparent Oral Volume of Distribution (Vz/F) Following Administration of DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48 and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Liters | 15.3369 (13.8) | 14.2222 (15.0) | 14.9889 (19.1)

13. Secondary Outcome: Concentration at 24hours Post-dose (C24) Following Administration of DTG
Description: as for outcome 2
Time Frame: 24 hours
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Micrograms per milliliter | 0.1763 (28.5) | 0.2167 (21.7) | 0.1917 (22.7)

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP was measured in a supine position after at least 5 minutes of rest for the participant in a quiet setting without any distractions using a completely automated device. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specific time point value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. All participants who were randomized and received at least one dose of study medication were part of Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 21
Millimeters of mercury
  SBP, Day 4 | 0.3 (10.50) | 4.9 (10.97) | 7.3 (9.59)
  DBP, Day 4 | -0.7 (6.83) | 1.8 (6.07) | 7.8 (7.05)

15. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in a supine position after at least 5 minutes of rest for the participant in a quiet setting without any distractions using a completely automated device. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specific time point value.
Time Frame: Baseline (Day -1) and Day 4
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 21
Beats per minute | 6.1 (11.06) | 6.8 (8.54) | 4.1 (11.38)

16. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose results in death,is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, any other situation according to medical or scientific judgement.
Time Frame: Up to Week 11
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 19 | 22
Participants
  Non-serious AEs | 3 | 3 | 4
  SAEs | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Hematology Parameters
Description: Blood samples were collected to analyze the following hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, hemoglobin, hematocrit, mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), percentage reticulocytes and red blood cell count. Data for clinically significant abnormal hematology parameters have been presented. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Baseline (Day -1)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 19 | 22
Participants | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Chemistry Parameters
Description: Blood samples were collected to analyze the following clinical chemistry parameters: Potassium, calcium, sodium, creatinine, glucose, alkaline phosphatase, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Blood urea nitrogen (BUN), total and direct bilirubin, total protein and creatine kinase. Data for clinically significant abnormal clinical chemistry parameters have been presented. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Baseline (Day -1)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 19 | 22
Participants | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Urine Parameters
Description: Urine samples were collected to analyze the following urinalysis parameters: specific gravity, potential of hydrogen (pH). Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Baseline (Day -1)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 19 | 22
Participants | 0 | 0 | 0

20. Primary Outcome: AUC From Time Zero to Infinity (AUC[0-inf]) for DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Hours*micrograms per milliliter | 12.8297 (23.0) | 14.8099 (21.8) | 13.0715 (23.8)
Statistical Analysis 1: Comparison: Prototype A vs DTG Reference; Test type: Equivalence — Bioequivalence is established when the 90% confidence interval of the ratio for AUC (0 to inf) between treatment formulations (Prototype A versus DTG Reference Treatment) are within the range of 0.80 to 1.25; Ratio = 0.96, 90% CI 2-sided [0.91 to 1.03]
Statistical Analysis 2: Comparison: Prototype B vs DTG Reference; Test type: Equivalence — Bioequivalence is established when the 90% confidence interval of the ratio for AUC (0 to inf) between treatment formulations (Prototype B versus DTG Reference Treatment) are within the range of 0.80 to 1.25; Ratio = 1.13, 90% CI [1.06 to 1.20]

21. Primary Outcome: Maximum Observed Concentration (Cmax) for DTG
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3,3.5, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Prototype A | Prototype B | DTG Reference
Number analyzed (Participants) | 18 | 18 | 22
Micrograms per milliliter | 0.9200 (14.4) | 0.9993 (17.6) | 0.8200 (26.1)
Statistical Analysis 1: Comparison: Prototype A vs DTG Reference; Test type: Equivalence — Bioequivalence is established when the 90% confidence interval of the ratio for Cmax between treatment formulations (Prototype A versus DTG Reference Treatment) are within the range of 0.80 to 1.25; Ratio = 1.09, 90% CI 2-sided [1.01 to 1.19]
Statistical Analysis 2: Comparison: Prototype B vs DTG Reference; Test type: Equivalence — Bioequivalence is established when the 90% confidence interval of the ratio for Cmax between treatment formulations (Prototype B versus DTG Reference Treatment) are within the range of 0.80 to 1.25; Ratio = 1.22, 90% CI 2-sided [1.13 to 1.33]

ADVERSE EVENTS:
Time Frame: Non-serious and serious adverse events were collected up to Week 11
Description: Non-serious AEs and SAEs were collected in the Safety Population
Arm/Group | Prototype A | Prototype B | DTG Reference
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 3/18 | 3/19 | 4/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prototype A (N=18) | Prototype B (N=19) | DTG Reference (N=22)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT03921723/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT03921723/SAP_001.pdf